CLINICAL TRIAL: NCT01937364
Title: Preventing Alcohol Withdrawal With Oral Baclofen: A Randomized, Placebo Controlled Trial
Brief Title: Preventing Alcohol Withdrawal With Oral Baclofen
Acronym: BACLOFEN III
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The enrollment in the study was too limited for meaningful data analysis.
Sponsor: Essentia Health (Other)
Responsible Party: Principal Investigator, Jeffrey E Lyon, MD, Essentia Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EIRH-13-1134
Record Dates: First submitted 2013-09-04; First posted 2013-09-09 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-03

CONDITIONS: Alcoholism; Alcohol Withdrawal
MeSH Terms: conditions — Alcoholism | interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo every eight hours as inpatients for 72 hours or until discharge if less than 72 hours.
  Interventions: Drug: Placebo
- Baclofen (Active Comparator): Baclofen 10 mg every 8 hours for 72 hours (9 doses) as an inpatient, or until discharge if before 72 hours.
  Interventions: Drug: Baclofen

INTERVENTIONS:
Drug: Baclofen — Baclofen 10 mg every 8 hours for 72 hours (9 doses) as an inpatient, or until discharge if before 72 hours.
  Other Names: lioresal
  Arms: Baclofen
Drug: Placebo — Identical appearing placebo every 8 hours for 72 hours (9 doses) as an inpatient, or until discharge if before 72 hours.
  Arms: Placebo

SUMMARY:
The purpose of this study is determine if the medication baclofen can prevent the symptoms of Alcohol Withdrawal Syndrome (AWS) in hospitalized patients who may be at risk for AWS. This medication is most often used for patients who have spasticity of their muscles due to a neuromuscular disease. In several European studies, and in an earlier study at Essentia Health (NCT00597701), baclofen has been found to have a significant effect on the severity of symptoms of AWS.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>21) admitted to inpatients units of 1 of 3 Essentia Health hospitals
* Patient placed on AWS watch protocol by admitting physicians.

Exclusion Criteria:

* Unable to provide informed consent
* Unable to take swallow oral medications (tube-fed patients are to be excluded)
* Admitted for AWS or with Clinical Institute Withdrawal Assessment of Alcohol Scale, Revised (CIWA-Ar) score >8 at baseline
* No alcohol intake for ≥ 48 hours or AUDIT score <12 at baseline
* Baclofen use at baseline
* Baclofen sensitivity
* Hospital discharge anticipated in within 48 hours
* Pregnant or breast feeding (urine pregnancy test required of women of child-bearing potential)
* Other active drug dependence (except tobacco)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey E Lyon, MD, Principal Investigator — Essentia Health
Locations (2):
- United States (2):
  - St. Mary's Medical Center, Duluth, Minnesota
  - Essentia Health Innovis Hospital, Fargo, North Dakota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Baclofen
Started | 9 | 8
Completed | 7 | 7
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Baclofen | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (11.37) | 48.9 (11.97) | 51.5 (11.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 7 | 7 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17
Baseline Clinical Institute Withdrawal Assessment of Alcohol Scale, Revised (CIWA-Ar) [Mean (Standard Deviation); unit: units on a scale] — Range: 0 to 67; larger values indicate greater severity
  units on a scale | 4.4 (2.01) | 3.9 (2.42) | 4.2 (2.16)

OUTCOME MEASURES:

1. Primary Outcome: Moderate or Severe Alcohol Withdrawal Syndrome
Description: Moderate or severe AWS was defined as a CIWA-AR score of at least 11.
Time Frame: 72 hours
Population: Subjects who either had AWS prior to the collection of the 72-hour CIWA-Ar score or had a CIWA-Ar score either recorded as the 72-hour CIWA-Ar score or occurring within the one-hour window for the 72-hour CIWA-Ar score are evaluable for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Baclofen
Number analyzed (Participants) | 5 | 7
Participants | 2 | 0
Statistical Analysis 1: Comparison: Placebo vs Baclofen; Test type: Superiority or Other; p = 0.0334, z-statistic with pooled estimate — One-sided p-value; Risk Difference (RD) = -0.40, 90% CI 2-sided [-0.7275 to -0.0206] — RD = Baclofen - Placebo

2. Secondary Outcome: Severity of Alcohol Withdrawal Symptoms as Measured on the CIWA-Ar Scale and Assessed at 24, 48, and 72 Hours After Enrollment
Description: Range: 0 to 67; larger values indicate greater severity
Time Frame: 72 hours
Population: All CIWA-Ar scores collected at and after the baseline measurement.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Baclofen
Number analyzed (Participants) | 9 | 8
units on a scale
  24 hours | 3.1325 (0.5283) | 2.4418 (0.5572)
  48 hours | 1.7913 (0.4666) | 1.9878 (0.4430)
  72 hours | 0.4501 (0.5646) | 1.5339 (0.4179)
Statistical Analysis 1: Comparison: Placebo vs Baclofen; Baclofen - Placebo; 24 hours; Test type: Superiority or Other; p = 0.3744, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo vs Baclofen; Baclofen - Placebo; 48 hours; Test type: Superiority or Other; p = 0.7616, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo vs Baclofen; Baclofen - Placebo; 72 hours; Test type: Superiority or Other; p = 0.1393, Mixed Models Analysis

3. Secondary Outcome: Peak and Total Benzodiazepine Dose Required
Time Frame: 72 hours
Measure: Median (Inter-Quartile Range); unit: Doses
Arm/Group | Placebo | Baclofen
Number analyzed (Participants) | 9 | 8
Doses
  Peak Ativan 1mg PO equivalent dose | 1.0 [0.0 to 2.0] | 0.5 [0.0 to 1.0]
  Total Ativan 1mg PO equivalent dose | 1.0 [0.0 to 3.0] | 0.5 [0.0 to 2.5]
Statistical Analysis 1: Comparison: Placebo vs Baclofen; Test type: Superiority or Other; p = 0.33, Wilcoxon (Mann-Whitney) — Baclofen - Placebo; Peak Ativan 1mg PO equivalent dose
Statistical Analysis 2: Comparison: Placebo vs Baclofen; Baclofen - Placebo; Total Ativan 1mg PO equivalent dose; Test type: Superiority or Other; p = 0.80, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Placebo | Baclofen
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes